CLINICAL TRIAL: NCT07238257
Title: Effectiveness of Digital Health Interventions on Community Health Care Among Middle-aged and Elderly Population in Taiwan: 6-month Cluster Randomized Trial
Brief Title: Effectiveness of Digital Health Intervention on Community Health Care in Middle-aged and Older Population in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202201534B0
Record Dates: First submitted 2025-10-01; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Hypertension (HTN); Type 2 Diabetes Mellitus (T2DM); Hyperuricemia; Hypercholesterolemia and Hyperlipidemia; Overweight (BMI > 25); Sleep Quality; Health Promotion
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Hyperuricemia; Hypercholesterolemia; Hyperlipidemias; Overweight; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Digital Health Program) (Experimental): Participants in this arm used smart devices to measure physiological data, including blood pressure, blood glucose, uric acid, cholesterol, and electrocardiograms. The data were automatically uploaded to a cloud-based health management platform. Physicians reviewed the data monthly and provided personalized consultations and health education during the 6-month intervention period.
  Interventions: Device: Digital Health Program with Smart Devices
- Control Group - Usual Care (No Intervention): Participants in this arm received usual community health care and did not use smart devices or the digital health management platform. No additional physician consultations or structured health education sessions were provided beyond the standard community health services.

INTERVENTIONS:
Device: Digital Health Program with Smart Devices — Participants in the intervention group used smart devices to measure physiological parameters, including blood pressure, blood glucose, uric acid, cholesterol, and electrocardiograms. These data were automatically uploaded to a cloud-based health management platform. Physicians reviewed the data monthly and provided personalized consultations and health education for 6 months.
  Arms: Intervention Group (Digital Health Program)

SUMMARY:
This study aims to evaluate the effectiveness of a digital health intervention for community-dwelling middle-aged and older adults in Taiwan. A total of 199 participants from four randomly selected communities will be enrolled in a 6-month cluster randomized trial. Participants in the intervention group will use smart devices to record physiological data, which are automatically uploaded to a cloud-based health management platform. Physicians will review the data monthly and provide personalized consultations and health education. Primary outcomes include anthropometric measures, biochemical indices, electrocardiograms, and self-reported health and sleep quality.

DETAILED DESCRIPTION:
This 6-month cluster randomized trial is conducted in Guishan District, Taoyuan City, Taiwan, to examine the impact of a digital health intervention on community health outcomes among adults aged 50 years and older.

From 32 eligible communities, four are randomly selected. Participants must have resided in the community for at least six months, be aged 50 years or older, and provide informed consent. Individuals with severe cognitive impairment, terminal illness, or an inability to use basic digital devices are excluded.

Participants in the intervention group will use smart devices to measure blood pressure, fasting glucose, uric acid, total cholesterol, and electrocardiograms. The data are automatically synchronized with a cloud-based health management platform. Physicians will review data monthly and provide individualized consultations and health education sessions at baseline, 3 months, and 6 months.

Primary outcomes include anthropometric indices (BMI, body fat percentage, visceral fat rating, skeletal muscle mass index), biochemical markers (fasting glucose, uric acid, cholesterol), and self-reported health and sleep quality. Secondary outcomes include trends in physiological indicators and associations among cardiometabolic risk factors.

Ethical approval was obtained from the Institutional Review Board of Chang Gung Memorial Hospital (IRB No.: 202201534B0). Written informed consent is obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 years and older
* Resided in the community for at least 6 months
* Able and willing to provide written informed consent

Exclusion Criteria:

* Severe cognitive impairment
* Terminal illness
* Inability to operate basic digital devices (e.g., smartphone, health monitoring device)
* Declined to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Blood Glucose | Baseline, 3 months, 6 months
  Measurement: Laboratory glucose value in milligrams per deciliter (mg/dL). Range: Typically 50-500 mg/dL observed in human plasma. Directionality: Higher values indicate worse glycemic control. Abnormal thresholds: FPG ≥ 100 mg/dL or PPG ≥ 140 mg/dL (American Diabetes Association criteria).
Change in Blood Pressure (Systolic and Diastolic) | Baseline, 3 months, 6 months
  Measurement: Systolic (mmHg) and diastolic (mmHg). Range: 70-250 mmHg (SBP); 40-150 mmHg (DBP). Directionality: Higher values indicate worse blood-pressure control. Abnormal threshold: SBP ≥ 130 mmHg or DBP ≥ 80 mmHg (2017 ACC/AHA guideline).
Change in Serum Uric Acid | Baseline, 3 months, 6 months
  Measurement: Serum uric-acid concentration (mg/dL). Range: 2-12 mg/dL. Directionality: Higher values indicate worse metabolic status. Abnormal threshold: > 7.0 mg/dL.
Change in Body Mass Index (BMI) | Baseline, 3 months, 6 months
  Measurement: Weight (kg) / height² (m²). Range: 10-60 kg/m². Directionality: Higher values indicate greater adiposity. Abnormal threshold: ≥ 24 kg/m² (Taiwanese overweight criterion).

SECONDARY OUTCOMES:
Change in Body Fat Percentage | Baseline, 3 months, 6 months
  Measurement range: 5-60 %. Directionality: Higher values indicate worse body-composition status. Abnormal threshold: ≥ 25 % (men) or ≥ 30 % (women).
Change in Visceral Fat Rating | Baseline, 3 months, 6 months
  Scale range: 1-59 points. Directionality: Higher scores indicate worse (greater) visceral-fat accumulation.
  Abnormal threshold: ≥ 10 points.
Change in Skeletal Muscle Mass Index (ASMI) | Baseline, 3 months, 6 months
  Measurement: Skeletal-muscle mass / height² (kg/m²). Typical range: 4.0-10.0 kg/m². Directionality: Higher values indicate better muscle mass. Cut-offs (AWGS 2019): < 7.0 kg/m² (men) or < 5.7 kg/m² (women) = low muscle mass.
Change in Self-Rated Health Status | Baseline, 3 months, 6 months
  Scale title: Self-Rated Health Scale (single-item global health question). Scale range: 1 = Excellent, 2 = Good, 3 = Fair, 4 = Poor, 5 = Very Poor. Directionality: Higher scores indicate worse perceived overall health.
Change in Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline, 3 months, 6 months
  Scale title: Pittsburgh Sleep Quality Index (PSQI), 19-item standardized questionnaire evaluating sleep over the previous month.
  Scale range: 0-21 points. Directionality: Higher scores indicate worse sleep quality. Interpretation: Total score > 5 = poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We have not made a final decision on sharing individual participant data (IPD). Data sharing will depend on institutional policies and participant privacy considerations.